CLINICAL TRIAL: NCT04685122
Title: Study of Subluxation Lens Biometrics and Postoperative Intraocular Lens Stability
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: xuwen2020-971
Record Dates: First submitted 2020-12-16; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Subluxation of Lens
MeSH Terms: conditions — Lens Subluxation | interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Phacoemulsification and intraocular lens implantation for cataract — Phacoemulsification and intraocular lens implantation for cataract

SUMMARY:
To compare the accuracy of four lens diameter measurement methods and to study the influencing factors of intraocular lens deviation after operation

ELIGIBILITY:
Inclusion Criteria:

(1) Subluxation of the lens is less than 180 degrees; (2) Part of the edge of the lens can be seen in the pupil area after the pupil is dilated

Exclusion Criteria:

(1) Total dislocation of the lens to the vitreous cavity (2) Patients with small eyeballs and small eyelid fissures (3) Patients younger than 18 years old (4) Congenital cataracts in both eyes (5) Corneal dystrophy or endothelial cell insufficiency (6) Chronic uvea Inflammation (7) Progressive fundus disease (8) Fragile capsular bag (9) Retinitis pigmentosa or pseudocapsular exfoliation syndrome

Ages: 20 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People whose subluxation of the lens is less than 180 degrees
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Lens diameter | through study completion, an average of 1 year
  Measured by related instruments before surgery and calculated by the circumference of the tension ring in the surgical video screenshot
The eccentric distance of the intraocular lens | 1 week postoperation
  The distance between the center of the lens plane and the center of the pupil plane is the eccentric distance of the lens.
The eccentric distance of the intraocular lens | 1 month postoperation
  The distance between the center of the lens plane and the center of the pupil plane is the eccentric distance of the lens.
The eccentric distance of the intraocular lens | 3 month postoperation
  The distance between the center of the lens plane and the center of the pupil plane is the eccentric distance of the lens.
The tilt angle of the intraocular lens | 1 week postoperation
  The angle between the plane of the lens and the plane of the pupil is the inclination of the lens
The tilt angle of the intraocular lens | 1 month postoperation
  The angle between the plane of the lens and the plane of the pupil is the inclination of the lens
The tilt angle of the intraocular lens | 3 month postoperation
  The angle between the plane of the lens and the plane of the pupil is the inclination of the lens

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No